CLINICAL TRIAL: NCT00947141
Title: Determining a Viral Load Threshold for Pre-emptive Therapy for Cytomegalovirus Infection in Transplant Patients Using Real Time Polymerase Chain Reaction (PCR) Monitoring
Brief Title: Determining a Viral Load Threshold for Treating Cytomegalovirus (CMV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6077; REC # 6077 (Other: NRES London - Central REC); Royal Free R and D # 5219 (Other: R&D department); ISRCTN03307563 (Other: ISRCTN)
Record Dates: First submitted 2009-06-12; First posted 2009-07-27 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Viraemia
Keywords: Optimising treatment of cytomegalovirus infection
MeSH Terms: conditions — Viremia | interventions — Ganciclovir; Valganciclovir; Foscarnet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Group A: (low level infection) has 2 arms:
  1. Start treatment when 2 consecutive levels CMV PCR >200copies / ml
  2. Monitor (Treatment starts when CMV PCR >3,000 copies / ml (current site clinical protocol))
  Interventions: Drug: ganciclovir (start when CMV PCR >200copies / ml x2); Other: Monitor (Treatment starts when CMV PCR >3,000 copies / ml)
- Group B (Experimental): Group B: (patients receiving pre-emptive therapy) has 2 arms:
  1. Stop treatment when 2 levels CMV PCR <3,000 copies / ml
  2. Monitor (Treatment stops when there are 2 consecutive levels of CMV PCR <200 copies / ml (current site clinical protocol))
  Interventions: Drug: Stop treatment when 2 levels CMV PCR <3,000 copies / ml; Other: Monitor (Treatment stops CMV PCR <200 copies / ml x2)

INTERVENTIONS:
Drug: ganciclovir (start when CMV PCR >200copies / ml x2) — Group A: Start ganciclovir when CMV PCR >200copies / ml x 2) . Participants are randomised to either Monitor or Treat. If monitored, treatment will only begin if viral load has increased > 3,000. If treated (and monitored) treat until <200 copies on 2 consecutive occasions.
  Routine standard of care would include treatment of Valganciclovir 900mg Tablet BD (dose adjusted for renal impairment), Ganciclovir 5mg/kg BD IV, or Foscarnet 60mg/kg according to randomisation within Group A or Group B
  Other Names: valganciclovir; foscarnet
  Arms: Group A
Other: Monitor (Treatment starts when CMV PCR >3,000 copies / ml) — Group A: CMV viral load between 200-3,000 copies/ml (on 2 occasions). Participants are randomised to either Monitor or Treat. If monitored, treatment will only begin if viral load has increased > 3,000. If treated (and monitored) treat until <200 copies on 2 consecutive occasions.
  Routine standard of care would include treatment of Valganciclovir 900mg Tablet BD (dose adjusted for renal impairment), Ganciclovir 5mg/kg BD IV, or Foscarnet 60mg/kg according to randomisation within Group A or Group B
  Other Names: valganciclovir; foscarnet
  Arms: Group A
Drug: Stop treatment when 2 levels CMV PCR <3,000 copies / ml — Group B: Viral load > 3,000 copies/ml. Participants are randomised to treat until < 3,000 copies/ml on 2 occasions or treat until <200 copies/ml on 2 consecutive occasions.
  Routine standard of care would include treatment of Valganciclovir 900mg Tablet BD (dose adjusted for renal impairment), Ganciclovir 5mg/kg BD IV, or Foscarnet 60mg/kg according to randomisation within Group A or Group B
  Other Names: valganciclovir; foscarnet
  Arms: Group B
Other: Monitor (Treatment stops CMV PCR <200 copies / ml x2) — Group B: Viral load > 3,000 copies/ml. Participants are randomised to treat until < 3,000 copies/ml on 2 occasions or treat until <200 copies/ml on 2 consecutive occasions.
  Routine standard of care would include treatment of Valganciclovir 900mg Tablet BD (dose adjusted for renal impairment), Ganciclovir 5mg/kg BD IV, or Foscarnet 60mg/kg according to randomisation within Group A or Group B
  Other Names: valganciclovir; foscarnet
  Arms: Group B

SUMMARY:
This study aims to determine: a) whether those patients with 'low level' viral load results (between 200 and 3,000 copies/ml) could be monitored as opposed to starting preemptive therapy with valganciclovir, ganciclovir and/or foscarnet; b) whether those patients with 'high level' viral load results (above 3,000 copies/ml) could stop preemptive therapy earlier, thus maximising the benefits of therapy and minimising its risks.

DETAILED DESCRIPTION:
Background and Study Rationale

In transplant recipients with CMV infection, the risk of developing CMV disease is directly proportional to the CMV DNA viral load. Historically at The Royal Free, Hampstead, patients were given preemptive therapy on the basis of two consecutive positive CMV PCR results as detected by a qualitative PCR technique. With the introduction of real time PCR, using a Taqman probe and the ABI7700 thermal cycler, it is possible to obtain rapid and sensitive results of viral load on clinical samples with a lower limit of detection of 200 copies/ml. Thus, viral load data can be incorporated into the clinical management of the patient.

From our natural history data, it has been shown that patients with CMV disease had a CMV PCR load ranging from 14,000 to 203 million (median 175,500). The lower bound of the 95% confidence limits of this distribution was 37,000 copies/ml and we aimed to initiate therapy in time to prevent CMV viral load reaching this value. To give a margin of safety, bearing in mind the 1 day average doubling-time of CMV and the timing of sampling twice-weekly, we therefore recommended that preemptive therapy be given once the viral load increases above 3,000 copies/ml. In the past, all patients with a CMV PCR load between 200 and 3,000 copies/ml have received preemptive treatment because the previous PCR assay did not give a quantitative result. As treatment is associated with side effects such as neutropaenia (ganciclovir) and renal impairment (foscarnet) it would be preferable to avoid unnecessary exposure where possible. This study aims to determine: a) whether those patients with 'low level' viral load results (between 200 and 3,000 copies/ml) could be monitored as opposed to starting preemptive therapy with valganciclovir, ganciclovir and/or foscarnet; b) whether those patients with 'high level' viral load results (above 3,000 copies/ml) could stop preemptive therapy earlier, thus maximising the benefits of therapy and minimising its risks.

Objectives

Primary Objectives

1. To define the number of patients in Group A with a low level of CMV reactivation who subsequently develop a viral load greater than 3000 copies/ml.
2. To define the number of patients in Group B who develop a second episode of a viral load above 3000 copies/ml after therapy has been discontinued at the defined viral load cut-offs.

Secondary Objectives

1. To define the duration of antiviral therapy needed to treat CMV viraemia.
2. To record the rate of increase in viral load prior to starting preemptive therapy.
3. To correlate viral loads with CMV specific immune function.

ELIGIBILITY:
Inclusion Criteria:

1. All Stem Cell, Renal and Liver Transplant recipients.
2. Willing to give informed consent.
3. For Group A) All patients with CMV viraemia (between 200 and 3000 copies/ml) in the liver, renal and stem cell groups in two consecutive samples & for Group B) Those patients requiring pre-emptive therapy because viral load is > 3,000 copies/ml.
4. All patients in either section of the study must be available for CMV PCR monitoring at least twice per week.

Exclusion Criteria:

1. Exclusion Criteria
2. Profound neutropaenia considered to preclude administration of ganciclovir or profound renal failure considered to preclude administration of foscarnet.
3. Inability to give informed consent.
4. In the stem cell group, Donor negative, Recipient negative transplants.
5. In the stem cell group: matched unrelated donors who are CMV seronegative.
6. Those patients who have been in Group A cannot then enter the Group B part. of the study. 5.2.6 Those patients who have been in Group B cannot then enter the Group A part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2003-02; Primary Completion 2011-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Group A # with low level of CMV who develop a viral load > 3000 copies/ml & Group B # who develop a 2nd episode of a viral load above 3000 copies/ml after therapy stopped. | At study completion

SECONDARY OUTCOMES:
To define the duration of antiviral therapy needed to treat CMV viraemia. To record the rate of increase in viral load prior to starting preemptive therapy & to correlate viral loads with CMV specific immune function. | At study completion

CONTACTS AND LOCATIONS:
Overall Officials: Professor Paul D Griffiths, MD DSc, Principal Investigator — University College, London
Locations (1):
- Royal Free London NHS Foundation Trust, Royal Free Hospital, Pond Street, London, United Kingdom

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045